CLINICAL TRIAL: NCT05907811
Title: The Effect of General Anesthesia and General Anesthesia Combined With Thoracic Epidural Anesthesia on Neuromuscular Block
Brief Title: General Anesthesia and General Anesthesia Combined With Thoracic Epidural Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Arzu Esen Tekeli, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2023/5
Record Dates: First submitted 2023-05-23; First posted 2023-06-18 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Thoracal Epidural Block
MeSH Terms: interventions — Blood Pressure; Heart Rate

STUDY DESIGN:
Intervention Model Description: Randomized prospective, controlled study
Who Masked: Participant, Outcomes Assessor
Masking Description: The cases were divided into 2 groups by the envelope method, and 30 subjects were included in the general anesthesia group (GA), and 30 subjects were included in the general anesthesia and thoracic epidural anesthesia group (GAE).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group general anesthesia (GA) (Sham Comparator): Anesthesia induction was applied to all patients with 1mg/kg lidocaine, 1μcg/kg fentanyl, 2mg/kg propofol, 0.6mg/kg rocuronium. When the TOF value was 0, the patients were intubated with an endotracheal tube. In the maintenance, desflurane at 8% concentration was used in a mixture of 50% O2 + 50% air. The time to reach 25% of the TOF value was noted in both groups. 0.1mg/kg rocuronium will be added to patients who reach 0.25.It was planned to administer 0.05mg/kg morphine 30 minutes before the end of the operation to the GA group.
  Interventions: Procedure: Neuromuscular blocker usage
- Group General anesthesia and Thoracal epidural (GAE) (Experimental): Electrodes were placed for TOF monitoring after thoracic epidural catheterization in the GAE group. Anesthesia induction was applied to all patients with 1mg/kg lidocaine, 1μcg/kg fentanyl, 2mg/kg propofol, 0.6mg/kg rocuronium. When the TOF value was 0, the patients were intubated with an endotracheal tube. In the maintenance, desflurane at 8% concentration was used in a mixture of 50% O2 + 50% air. The time to reach 25% of the TOF value was noted in both groups. 0.1mg/kg rocuronium will be added to patients who reach 0.25.The number of additional muscle relaxant requirements made will be recorded. In the GAE group, 5 ml of epidural medication will be given per hour. When the TOF value reached 70%, inhaler anesthetics were discontinued and the patients with a TOF value of 90% were extubated.
  Interventions: Procedure: Neuromuscular blocker usage

INTERVENTIONS:
Procedure: Neuromuscular blocker usage — The patients were followed up, the total amount of muscle relaxant used was determined, intraoperative effects and postoperative analgesic usage
  Other Names: Train of four (TOF); Blood pressure; Heart rate; Oksygen saturation; Visual analog scale

SUMMARY:
It was aimed to investigate whether epidural anesthesia added to general anesthesia has an effect on neuromuscular block.

DETAILED DESCRIPTION:
The study was carried out with patients who were evaluated preoperatively in the Department of Anesthesiology and Reanimation, Department of Anesthesiology, Faculty of Medicine, Yuzuncu Yıl University. Sixty ASA I-II group patients, aged between 18-65 and scheduled for gastric ca operation, were included in the study. Severe heart, lung, liver disease, kidney failure, bleeding diathesis, fever, infection, allergy to drugs to be used, those who refused to participate in the study, patients with hypothermic and acid-base disorders, electrolyte disorders such as hypokalemia, hypocalcemia, antibiotics, anticonvulsants, Those taking antiarrhythmic and cholinesterase inhibitors were excluded from the study.

The cases were divided into 2 groups by the envelope method, 30 people will be included in the general anesthesia group (GA), and 30 people will be included in the general anesthesia and thoracic epidural anesthesia group (GAE). After the patients who did not receive premedication were taken to the operating room, standard monitoring was provided with ECG, non-invasive arterial pressure, peripheral oxygen saturation. Peripheral vein cannulation was performed with a 20 gauge i.v. catheter, and a 4 mL/kg 0.9% NaCl infusion was started. In Group GAE, after preoperative asepsis was achieved, cutaneous-subcutaneous local anesthetic was infiltrated through the T7-9 space. The epidural space was determined by the loss of resistance method with a 16 gauge Tuohy epidural needle, and an 18 gauge epidural catheter was placed in the epidural space at a 4 cm angle in the cranial direction. The location of the catheter was confirmed by applying a test dose of 3 mL 2% lidocaine containing 5μ/ml adrenaline. After 5 minutes, 5 ml of 0.125% bupivacaine was given and the patient was placed in the supine position immediately afterwards. Electrodes were placed for TOF monitoring after thoracic epidural catheterization in the GAE group. Anesthesia induction was applied to all patients with 1mg/kg lidocaine, 1μcg/kg fentanyl, 2mg/kg propofol, 0.6mg/kg rocuronium. When the Train of four (TOF) value was 0, patients were intubated with an endotracheal tube (7-7.5 endotracheal tube (ETT) for women, 8-8.5 ETT for men). In maintenance, desflurane at 8% concentration was applied in a mixture of 50% O2 + 50% air. The time to reach 25% of the TOF value for both groups was noted. 0.1mg/kg rocuronium was added to patients who reached 0.25. The number of additional muscle relaxant requirements was recorded. In the GAE group, 5 ml of epidural drug was given every hour. In the GA group, 0.05mg/kg morphine was given 30 minutes before the end of the operation. Considering the time it took for the TOF value to reach 70%, the inhaler anesthetics were terminated and the patients with a TOF value of 90% were extubated.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II group
* 60 patients
* 18-65 who were scheduled for gastric ca operation were included in the study.

Exclusion Criteria:

* severe heart, lung, liver disease,
* kidney failure,
* bleeding diathesis,
* fever,
* infection,
* allergy to drugs to be used,
* those who refused to participate in the study,
* patients with hypothermic and acid-base disorders,
* electrolyte disorders
* antibiotics,
* anticonvulsants, Those taking antiarrhythmic, cholinesterase inhibitors will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Neuromuscular agent | 30 minute
  Total neuromuscular consumption

CONTACTS AND LOCATIONS:
Overall Officials: School of Medicine Department of Anesthesiology and Reanimation, Study Chair — Yuzuncu Yil University
Locations (1):
- Arzu Esen Tekeli, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Personal data of participating patients will not be shared in any way.